CLINICAL TRIAL: NCT03626571
Title: Molecular Imaging in Infective Endocarditis Using Hybrid Positron Emission Tomography/Magnetic Resonance Imaging (PET/MR) and Computed Tomography (PET/CT)
Brief Title: PET/MR Imaging In Patients With Infective Endocarditis
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC17012
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Native valve infective endocarditis: Patients with infective endocarditis of native valves of the heart with no contraindications to MRI scanning.
  Interventions: Other: 18F-FDG
- Prosthetic endocarditis: Patients with endocarditis of prosthetic heart valves or device-related infections.
  Interventions: Other: 18F-FDG
- Non-infective post-operative: Patients who have recently undergone valve or device implantation with no evidence of post-operative infection.
  Interventions: Other: 18F-FDG

INTERVENTIONS:
Other: 18F-FDG — Hybrid 18F-FDG PET/MR or PET/CT imaging for observational diagnostic purposes.

SUMMARY:
PET scanning (positron emission tomography) is a well-established technique used to identify areas of interest within the body. It involves injecting a radioactive tracer which highlights abnormal areas. It has recently been combined with CT (computed tomography) and MRI (magnetic resonance imaging) scanning to more accurately identify abnormalities within the heart. Infective endocarditis (infection of the heart valves or lining of the heart) and device infection (where a pacemaker device or wire becomes infected) are of particular interest in this area.

The study makes use of hybrid PET/MR scanning using a designated scanner which enables PET scanning combined with MRI scanning. PET scanning combined with CT scanning will be used instead for patients who aren't able to undergo MRI scanning. This will allow abnormal areas within the heart in these conditions to be characterised, alongside treatment regimens, in a way which hasn't been done before.

All participants will undergo PET scanning, where a radioactive tracer is injected into a vein before the scan. The radioactive substance only lasts for a short time, passed out of the body in urine. Patients with infective endocarditis involving their own heart valve will undergo an MRI scan as part of the PET scan. Patients with infective endocarditis involving a metal or prosthetic heart valve and also patients who have pacemaker infections, instead of an MRI, will have a CT scan. The reason for this is that CT is better for looking at metal and prosthetic heart valves and patients with pacemakers can't have MRI scans because the strong magnet in the scanner can affect the pacemaker. The scan will be performed twice; once before treatment and once after treatment has been established.

If successful, this imaging method will play a key role in diagnosing, quantifying and monitoring these conditions.

ELIGIBILITY:
Inclusion Criteria:

Age criteria as follows:

* Native valve endocarditis >30 years
* Prosthetic valve endocarditis/device infection >50 years
* Non-infective post-operative patients >65 years

Additional inclusion criteria:

* Completion of informed consent
* Established diagnosis of one of the conditions listed below:

I. Native valve infective endocarditis; established diagnosis by Dukes criteria II. Prosthetic valve or device-related infection; established diagnosis by Dukes criteria (in the case of valves), or by microbiological, haematological and biochemical grounds (in the case of device-related infection) III. Recent implant of prosthetic valve and/or cardiac device

Exclusion Criteria:

* Inability or unwilling to give informed consent
* Women who are pregnant, breastfeeding or of child-bearing potential (women who have experienced menarche, are pre-menopausal and have not been sterilised) will not be enrolled into the trial
* Major intercurrent illness with life-expectancy <2 years
* Renal dysfunction (eGFR less than or equal to 30ml/min/1.73m2)
* Adverse reaction or hypersensitivity to 18F-FDG PET tracer
* NYHA Class IV heart failure
* Insulin-dependent diabetes mellitus
* Patients with atrial fibrillation and poor rate control
* Contraindications to MR for patients in the groups undergoing PET/MR including any patient with suspected metal in their eyes
* Previous history of contrast allergy of adverse reactions (iodinated contrast in patients undergoing PET/CT and gadolinium in patients undergoing PET/MR)

Min Age: 30 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients attending the Edinburgh Heart Centre will be invited to participate. Inpatients and outpatients are eligible. Healthy volunteers will be invited to participate by local recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Myocardial 18F-FDG uptake | 1 year
  Quantification of myocardial PET tracer uptake, early and late time-points

CONTACTS AND LOCATIONS:
Overall Officials: Marc R Dweck, MD PhD, Study Director — University of Edinburgh
Locations (1):
- Queen's Medical Research Institute, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No